CLINICAL TRIAL: NCT01856023
Title: Open-Label, Randomized, Multi-Center Study Comparing the Sequence of High Dose Aldesleukin (Interleukin-2) and Ipilimumab (Yervoy) in Patients With Metastatic Melanoma
Brief Title: HD IL-2 + Ipilimumab in Patients With Metastatic Melanoma
Acronym: PROCLIVITY02
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: slow accrual & early closure
Sponsor: Clinigen, Inc. (Industry)
Collaborators: M.D. Anderson Cancer Center (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 12PLK02
Record Dates: First submitted 2013-05-10; First posted 2013-05-17 (Estimated); Results first posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-03

CONDITIONS: Metastatic Melanoma
Keywords: melanoma; metastatic; skin cancer; Stage IV; interleukin-2
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis; Skin Neoplasms | interventions — Interleukin-2; aldesleukin; Interleukins; Ipilimumab

STUDY DESIGN:
Intervention Model Description: assess the sequenced use of HD IL2 and IPI in metastatic melanoma patients
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Arm 1 (Active Comparator): Patients will receive two courses (four cycles) of High Dose Interleukin-2 (HD IL-2) followed by one course (four doses) of ipilimumab.
  Interventions: Drug: High Dose Interleukin-2; Drug: Ipilimumab
- Treatment Arm 2 (Active Comparator): Patients will receive one course (four doses) of ipilimumab followed by two courses (four cycles) of HD IL-2.
  Interventions: Drug: High Dose Interleukin-2; Drug: Ipilimumab

INTERVENTIONS:
Drug: High Dose Interleukin-2
  Other Names: Aldesleukin; Proleukin; interleukin
Drug: Ipilimumab
  Other Names: Yervoy; anti-CTLA4

SUMMARY:
Phase IV, open-label, randomized, two-arm, multi-center study in patients with metastatic melanoma who are treatment naïve or have previously received a single non-immunologic therapy.

Treatment Arm 1: "HD IL-2 first, then ipilimumab" Patients will receive two courses (four cycles) of High Dose Interleukin-2 (HD IL-2) followed by one course (four doses) of ipilimumab.

Treatment Arm 2: Ipilimumab first then HD IL-2 Patients will receive one course (four doses) of ipilimumab followed by two courses (four cycles) of HD IL-2.

DETAILED DESCRIPTION:
All patients will receive IL-2 at 600,000 international units per kilogram (kg) by intravenous bolus (IVB) every 8 hours for up to 14 planned doses with an additional cycle 14 days after the first.

Ipilimumab 3mg/kg IV infusion Q3 weeks up to 4 doses4 doses A 3-6 week interval been the administration of the two drugs to allow for resolution of treatment-related toxicities.

If corticosteroids were required during Ipilimumab administration, a 2-week period from discontinuation of steroid treatment to start of HD IL-2.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years or older
* Confirmed and measurable metastatic melanoma with at least one measurable lesion for evaluation of response
* Meets the requirements for HD IL-2 therapy per Institutional guidelines
* Meets the requirements for ipilimumab therapy per Institutional guidelines
* Treatment naïve or has received only one systemic therapy apart from adjuvant therapy.
* At least 4 weeks since last adjuvant therapy or other cancer treatment
* Willing and able to give informed consent and participate in study procedures as described in the 12PLK02 and 10PLK13 protocols. Patients consented for 12PLK02 will also be asked to participate in the 10PLK13 PROCLAIM registry study.

Exclusion Criteria:

* Patients with known or suspected infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), hepatitis B virus (HBV) or other infectious hepatitis
* Pregnant, nursing or planning to become pregnant
* Untreated brain metastases. (Brain metastases that have been treated, which no longer require corticosteroid therapy and are without progression by MRI at least 6 weeks after definitive therapy are acceptable.)
* Received prior ipilimumab therapy (Prior Adjuvant Ipilimumab and Adjuvant Interferon are permitted with a minimum 4 week washout)
* Received prior HD IL-2 therapy.
* Received investigational drug within 30 days prior to study dosing. Patients may participate in non-interventional or observational clinical studies, including the 10PLK13 PROCLAIM registry study.
* Concomitant disease or condition that would interfere with the conduct of the study or that would, in the opinion of the Investigator, pose an unacceptable risk to the patient in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sapna Patel, MD, Principal Investigator — MD Anderson; William Sharfman, MD, Principal Investigator — Johns Hopkins University; James Lowder, MD, Principal Investigator — Prometheus Labs
Locations (12):
- United States (12):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - Moores UCSD Cancer Center, La Jolla, California
  - MSMC Research Program, Miami Beach, Florida
  - Oncology Specialists, SC, Park Ridge, Illinois
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Johns Hopkins Medicine, Lutherville, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - Nebraska Cancer Specialists, Midwest Cancer Center - Legacy, Omaha, Nebraska
  - Columbia University Medical Center, Herbert Irving Comprehensive Cancer Center, New York, New York
  - Duke University Health System, Durham, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - MD Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study initiation Sept 11, 2013 - Early Study Termination August 18, 2015 Planned accrual 50 pts/ arm.
Pre-assignment Details: Patients will be randomized to receive both treatments in different sequence: Arm 1 IL-2 followed by Ipi; Arm 2 IPI followed by IL-2 Evaluable Patients will have received at least 50% of dose of both study drugs and completed assessment; Safety Population are all patients who received 1 dose of either study drug; Intent to treat
Groups:
- Treatment Arm 1 HD IL-2 1st Followed by Ipilimumab: Patients will receive two courses (four cycles) of High Dose Interleukin-2 (HD IL-2) followed by one course (four doses) of ipilimumab.
  3-6 week interval between the two drugs to allow resolution of treatment-related toxicities.
  High Dose Interleukin-600,000IU/kg IV every 8 hours up to 14 doses per cycle
  Ipilimumab 3mg/kg IV every 3 weeks up to 4 doses
- Treatment Arm 2 Ipilimumab 1st Followed by HD IL-2: Patients will receive one course (four doses) of ipilimumab followed by two courses (four cycles) of HD IL-2.
  3-6 week interval between the two drugs to allow resolution of treatment-related toxicities.
  High Dose Interleukin-600,000IU/kg IV every 8 hours up to 14 doses per cycle
  Ipilimumab 3mg/kg IV every 3 weeks up to 4 doses
Period: Overall Study
Arm/Group | Treatment Arm 1 HD IL-2 1st Followed by Ipilimumab | Treatment Arm 2 Ipilimumab 1st Followed by HD IL-2
Started (I pt withdrew consent prior to receiving study drug- should have been listed as screen failure) | 13 | 16
Intent to Treat: Received One Dose of Study Drug | 12 | 16
Evaluable: Received 50% of Each Study Drug | 8 | 10
Completed (completed all study requirements) | 3 | 4
Not Completed | 10 | 12
Not completed — Death | 1 | 2
Not completed — Adverse Event | 2 | 1
Not completed — Lack of Efficacy | 5 | 5
Not completed — non compliance, study closure | 1 | 3
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment Arm 1 IL-2 First: Patients will receive two courses (four cycles) of High Dose Interleukin-2 (HD IL-2) followed by one course (four doses) of ipilimumab.
  High Dose Interleukin-2
  Ipilimumab
- Treatment Arm 2 Ipi First: Patients will receive one course (four doses) of ipilimumab followed by two courses (four cycles) of HD IL-2.
  High Dose Interleukin-2
  Ipilimumab
- Total: Total of all reporting groups
Arm/Group | Treatment Arm 1 IL-2 First | Treatment Arm 2 Ipi First | Total
Number analyzed (Participants) | 13 | 16 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 14 | 26
  >=65 years | 1 | 2 | 3
Age, Continuous [Median (Full Range); unit: years] | 49.5 [32 to 70] | 46 [20 to 69] | 48 [20 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 8 | 12 | 20
Region of Enrollment [Number; unit: participants]
  United States | 13 | 16 | 29

OUTCOME MEASURES:

1. Primary Outcome: Estimated One-year OS in the Evaluable Population in Each Treatment Arm Separately
Description: evaluable patients who received at least 50% of both research drugs and had their disease re-evaluated after baseline; defined in days for the start of the first treatment to death.
  percent of patients alive at 1 year; estimates were assessed using Kaplan-Meier method for the entire subject population for each treatment arm separately.
Time Frame: start of first treatment to date of death from any cause and patients alive at their last evaluation date were censored up to 1 year.
Population: patients who received at least 50% of both research drugs as planned-and had their disease re-evaluated after baseline; patients who exhibited PD or died before the end of one course of treatment were also considered evaluable
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Treatment Arm 1: Patients will receive 2 courses (four cycles) of High Dose Interleukin-2 (HD IL-2) followed by one course (four doses) of ipilimumab.
  3-6 week interval between the two drugs administered to resolve treatment-related toxicities
- Treatment Arm 2: Patients will receive one course (four doses) of ipilimumab followed by two courses (four cycles) of HD IL-2.
  3-6 week interval between the two drugs administered to resolve treatment-related toxicities
Arm/Group | Treatment Arm 1 | Treatment Arm 2
Number analyzed (Participants) | 8 | 10
percentage of participants | 73 [38 to 91] | 75 [40 to 92]
Statistical Analysis 1: Comparison: Treatment Arm 1 vs Treatment Arm 2; OS rates of the Evaluable population in entire cohort was compared with the historical control rate of 46% (Hodi, et al NEJM 2010) using a one-sample binomial test due to early termination of enrollment without reaching target accrual; planned analysis to be the difference between treatment arms using log-rank test. One year OS along with 95% CI estimated for entire population and each treatment arm separately; Test type: Superiority — one -sample binomial test - 1-year estimated OS for these 28 patients was 75% (95%CI: 51%, 88%); p = .001, Log Rank — compared to the historical control rate of 46% one year survival

2. Secondary Outcome: Progression-free Survival
Description: duration of time (in Days) from start of the first treatment to the time of objective disease progression or death at one year. The immune-related response criteria (irRC) determined based on tumor burden calculated on the WHO method of multiplying the perpendicular dimensions of all lesions are summed to obtain the tumor burden. The total tumor burden + SPD (index lesions) + SPD (new measurable lesions) Based on CT scans and Physical exam at designated timepoints. CR- Disappearance of all known disease; PR>/equal to decrease; SD Neither CR or PD; PD 25%increase; new lesion.
Time Frame: 5-11 weeks, 13-19 Weeks, 24-30 weeks and 1 year
Population: Evaluable patients who received up to 50% of the planned cycles of therapy in both study drugs; comparison of the sequences of therapy between treatment arms
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Treatment Arm 1 HD IL-2 1st Followed by Ipilimumab: Patients will receive two courses (four cycles) of High Dose Interleukin-2 (HD IL-2) followed by one course (four doses) of ipilimumab.
  High Dose Interleukin-600,000IU/kg IV every 8 hours up to 14 doses per cycle
  Ipilimumab 3mg/kg IV every 3 weeks up to 4 doses
- Treatment Arm 2 Ipilimumab 1st Followed by HD IL-2: Patients will receive one course (four doses) of ipilimumab followed by two courses (four cycles) of HD IL-2.
  High Dose Interleukin-2
  Ipilimumab
Arm/Group | Treatment Arm 1 HD IL-2 1st Followed by Ipilimumab | Treatment Arm 2 Ipilimumab 1st Followed by HD IL-2
Number analyzed (Participants) | 8 | 10
days | 58 [18 to 84] | 80 [41 to 95]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored/ assessed for up to 30 weeks after 1st dose of study drug. All -cause mortality monitored/assessed up to 1 year.
Description: AEs and SAEs listed as described below by arm and not specific for each drug. Adverse events were not assessed separately for each drug; However, side effects of each drug are established and commented in the final manuscript.
Groups:
- Treatment Arm 1 HD IL-2 Administered 1st Followed by Ipilimumab: Patients will receive two courses (four cycles) of High Dose Interleukin-2 (HD IL-2) followed by one course (four doses) of ipilimumab.
  3-6 week interval between the two drugs to allow resolution of treatment-related toxicities.
  High Dose Interleukin-600,000IU/kg IV every 8 hours up to 14 doses per cycle Ipilimumab 3mg/kg IV every 3 weeks up to 4 doses
- Treatment Arm 2 Ipilimumab Administered 1st Followed by HD IL-2: Patients will receive one course (four doses) of ipilimumab followed by two courses (four cycles) of HD IL-2.
  3-6 week interval between the two drugs to allow resolution of treatment-related toxicities.
  High Dose Interleukin-600,000IU/kg IV every 8 hours up to 14 doses per cycle Ipilimumab 3mg/kg IV every 3 weeks up to 4 doses
Arm/Group | Treatment Arm 1 HD IL-2 Administered 1st Followed by Ipilimumab | Treatment Arm 2 Ipilimumab Administered 1st Followed by HD IL-2
All-Cause Mortality (participants affected / at risk) | 1/13 | 2/16
Serious Adverse Events (participants affected / at risk) | 9/13 | 10/16
Other Adverse Events (participants affected / at risk) | 9/13 | 10/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm 1 HD IL-2 Administered 1st Followed by Ipilimumab (N=13) | Treatment Arm 2 Ipilimumab Administered 1st Followed by HD IL-2 (N=16)
Diarrhea (Gastrointestinal disorders) | 1 | 0
colitis (Gastrointestinal disorders) | 0 | 2
ascites (Gastrointestinal disorders) | 0 | 1
intestinal perforation (Gastrointestinal disorders) | 0 | 1
back pain, neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0
supraventricular tachycardia, ventricular tachycardia (Cardiac disorders) | 2 | 0
Autoimmune encephalitis, intracranial Hemorrhage (Nervous system disorders) | 2 | 0
Sedation, mental Status change (Psychiatric disorders) | 0 | 1 (2)
Pneumonia (Infections and infestations) | 0 | 2
Perihepatic Abscess (Infections and infestations) | 0 | 1
Respiratory Failure, Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
renal failure acute (Renal and urinary disorders) | 0 | 1
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 1
embolism (Vascular disorders) | 1 | 0
wound infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm 1 HD IL-2 Administered 1st Followed by Ipilimumab (N=13) | Treatment Arm 2 Ipilimumab Administered 1st Followed by HD IL-2 (N=16)
diarrhea (Gastrointestinal disorders) | 4 | 1
Back pain, neck pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Ascites (Metabolism and nutrition disorders) | 0 | 1
increased creatinine (Blood and lymphatic system disorders) | 3 | 0
increased ALT (Blood and lymphatic system disorders) | 1 | 1
Increased AST (Blood and lymphatic system disorders) | 1 | 1
Increased BUN (Blood and lymphatic system disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
Acute Kidney Injury (Renal and urinary disorders) | 8 | 2
Urinary Retention (Renal and urinary disorders) | 2 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3 | 0
Extremity Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Peripheral Edema (General disorders) | 3 | 1
Fatigue (General disorders) | 1 | 2
Hypotension (Vascular disorders) | 3 | 1
Flushing (Vascular disorders) | 3 | 0
Sinus Tachycardia (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 2
Metabolic Acidosis (Metabolism and nutrition disorders) | 2 | 0
Paresthesia (Nervous system disorders) | 0 | 2
Mental Status Change, Sedation (Psychiatric disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
This study enrollment planned for 50 in each arm; but ended early 29 pts enrolled due to change in treatment options; the purpose of the study was to determine which sequence of approved therapy was more effective and safe; this was not a planned cross-over study complete data collection and final summary is limited due to limited data available Due to sponsor changes, and databases are no longer available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No